CLINICAL TRIAL: NCT03793504
Title: Cardio-Respiratory Response of an Exercise Training Session With Ergocycle or Treadmill Compared to an Adapted Physical Activity Session on a Wii, in Patients With Pulmonary Disease
Brief Title: Cardio-Respiratory Response of a Training Session Versus an Adapted Physical Activity Session
Acronym: WIIRR
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: WIIRR (29BRC18.0250)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease
Keywords: pulmonary rehabilitation; exercise; physical activity
MeSH Terms: conditions — Lung Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of this study is to show that training session with nintendo WII requires the same cardiorespiratory demand than training session on ergocycle or treadmill, traditionally used in pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* patients with pulmonary disease

Exclusion Criteria:

* exacerbation of the pulmonary disease
* Weight >150Kg
* Refusal to participate
* People in pre and post surgical rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pulmonary disease admitted in pulmonary rehabilitation unit of CHU Brest
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
compare heart rate between a training session on cycle or treadmill and a training session on Nintendo WII | one day
  heart rate (pulse per minute) at the end of each session

SECONDARY OUTCOMES:
compare dyspnea between a training session on cycle or treadmill and a training session on nintendo WII | one day
  dyspnea (borg scale) at the end of each session
compare lower limb muscle fatigue between a training session on cycle or treadmill and a training session on nintendo WII | one day
  lower limb muscle fatigue (borg scale) at the end of each session
compare pulse oxymetry (SpO2) between a training session on cycle or treadmill and a training session on nintendo WII | one day
  SpO2 at the end of each session
Compare the felt pleasure between a training session on cycle or treadmill and a training session on nintendo WII | one day
  felt pleasure (likert scale) at the end of each session

CONTACTS AND LOCATIONS:
Overall Officials: Marc BEAUMONT, PhD, Principal Investigator — CHRU de Brest
Locations (1):
- CH Morlaix, Morlaix, France